CLINICAL TRIAL: NCT06315543
Title: Effect of Increased Daily Water Intake in Patients With Hyperuricemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20222255-F-1
Record Dates: First submitted 2024-02-18; First posted 2024-03-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-01

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adequate drinking water intervention group (Experimental): increase drinking water by 1650mL per day (3 bottles of 550mL bottled water) on the basis of original drinking water
  Interventions: Dietary Supplement: Drink water
- Water intake observation group (No Intervention): maintain original water intake

INTERVENTIONS:
Dietary Supplement: Drink water — Increase drinking water by 1650mL per day (3 bottles of 550mL bottled water)
  Arms: Adequate drinking water intervention group

SUMMARY:
The purpose of this study is to explore the clinical effect of reducing uric acid by drinking water, and provide scientific evidence and clinical guidance for reducing uric acid by drinking water. The study design was a multicenter, prospective, randomized controlled clinical trial with a total of 88 participants (Group A n=44; Group B n=44). 1. Inclusion criteria: patients with hyperuricemia (fasting uric acid between 420-540μmol/L twice on different days and no drug treatment); Aged 18-65 years; Less than 1500mL of daily water intake recommended by the minimum dietary guidelines (assessed by dietary review combined with water diaries); Fully informed consent. Sign informed consent. 2. Exclusion criteria: Patients with heart, liver and kidney insufficiency; Patients with severe or uncontrollable organic diseases that may interfere with the study parameters (such as tumors, cardiovascular, pulmonary and digestive diseases, hypertension, hyperlipidemia, hyperglycemia, thyroid diseases) or psychiatric disorders that affect eating behavior (such as primary polydipsia, bulimia nervosa, Psychiatric disorders, etc.); Patients with secondary hyperuricemia caused by other diseases; Patients who have taken any drug that causes changes in uric acid within five half-lives of the drug; Receiving treatment that can change the assessment of hydration status in the study (taking diuretics, glucocorticoids, or treatments that interfere with metabolism); Those who have gastrointestinal discomfort or a history of gastrointestinal surgery after drinking water, and other patients who are not suitable to drink too much water. A total of 88 subjects were included according to the exclusion criteria. The subjects were divided into two groups: Group A adequate drinking water intervention group (drinking an additional 1650mL of water per day (3 bottles of 550mL bottled water) on the basis of the original drinking water volume); Group B constant drinking water observation group (maintaining the original drinking water volume). During the 2-week observation period, the effects of sufficient drinking water on blood uric acid, urine osmotic pressure and other indicators were evaluated, and the effectiveness of sufficient drinking water in reducing blood uric acid was determined, and the applicable population was explored.

Observation items and detection time: 1. During the screening period, the following data were collected: age, nationality, place of residence, education, occupation, height, weight, waist circumference, disease history, drug use history, drinking, smoking, normal water intake, urine volume, urine color and uric acid value. 2. Pre-test data: drinking water, urination, diet, psychological investigation, blood uric acid, blood biochemistry, routine blood routine, urine routine, uric acid, urine osmotic pressure, systolic blood pressure, diastolic blood pressure, heart rate, frequency of gout attack, whether to take uric-lowering drugs, whether to take other drugs that affect uric acid. 3. After the test: Fasting blood uric acid was monitored on the 2nd, 4th, 6th, 8th, 10th and 14th day respectively; Urge patients to record water diary and urination diary every day. At the end of the experiment, blood uric acid, blood biochemistry, blood routine, urine routine, urine uric acid, urine osmotic pressure, systolic blood pressure, diastolic blood pressure and heart rate were tested again. Safety assessment indicators: edema, gastrointestinal discomfort, electrolytes, blood pressure, heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hyperuricemia (fasting uric acid values between 420-540μmol/L twice on different days and no drug treatment)
* Men between the ages of 18-65
* Daily water intake of less than 1500 mL recommended by the minimum dietary guidelines (assessed by dietary review combined with water diary)
* Fully informed consent, sign informed consent

Exclusion Criteria:

* Patients with heart, liver and kidney insufficiency.
* Patients with severe or uncontrollable organic diseases that may interfere with the study parameters (such as tumors, cardiovascular, pulmonary and digestive diseases, hypertension, hyperlipidemia, hyperglycemia, thyroid diseases) or psychiatric disorders that affect eating behavior (such as primary polydipsia, bulimia nervosa, Psychiatric disorders, etc.).
* Patients with secondary hyperuricemia caused by other diseases.
* Patients who have taken any drug that causes changes in uric acid within five half-lives of the drug.
* Receiving treatment that can change the assessment of hydration status in the study (taking diuretics, glucocorticoids, or treatments that interfere with metabolism).
* Those who have gastrointestinal discomfort or a history of gastrointestinal surgery after drinking water, and other patients who are not suitable to drink too much water.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Blood uric acid change | 2 weeks
  Changes of uric acid value after drinking water intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China